CLINICAL TRIAL: NCT02506192
Title: Gulf War Illness Inflammation Reduction Trial
Acronym: GWIIRT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ronald Bach, Research Health Scientist, Minneapolis Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4554-A
Record Dates: First submitted 2015-07-20; First posted 2015-07-23 (Estimated); Results first posted 2023-12-06 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Chronic Inflammation; Chronic Pain; Fatigue; Cognitive Impairment
Keywords: Gulf War Illness; Chronic Inflammation; Modified-Release Prednisone; Health-Related Quality of Life
MeSH Terms: conditions — Chronic Pain; Fatigue; Cognitive Dysfunction | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double-blind, placebo-controlled
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Modified-Release Prednisone (Experimental): Take oral tablets as directed (2x5mg) with food each evening at bedtime- approximately 10:00 pm
  Interventions: Drug: Modified-Release Prednisone
- Placebo (Placebo Comparator): Take oral tablets as directed (2x5mg) with food each evening at bedtime-approximately 10:00 pm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Modified-Release Prednisone — Modified-Release Prednisone oral tablets (2x5mg) daily for 8 weeks
  Other Names: Rayos
  Arms: Modified-Release Prednisone
Drug: Placebo — Placebo oral tablets (2x5mg) daily for 8 weeks
  Other Names: sugar pill, inactive substance
  Arms: Placebo

SUMMARY:
The primary objective of this clinical trial is to determine if treatment with an anti-inflammatory drug (delayed-release prednisone) improves the health-related quality of life (HRQOL) of veterans with Gulf War Illness (GWI). The primary outcome measure is a change from baseline of HRQOL with respect to physical functioning and symptoms. Secondary outcomes measures include changes from baseline levels of GWI-associated biomarkers of inflammation in peripheral blood, GWI-associated symptoms (chronic pain, fatigue, and cognitive impairment), and HRQOL with respect to mental functioning.

DETAILED DESCRIPTION:
During Desert Shield and Desert Storm (Aug 2, 1990 to July 31,1991) 696,841 United States Military personnel were deployed to the Kuwaiti Theater of Operations. Today approximately one-third of those veterans are suffering from GWI, an unexplained chronic multi-symptom illness. Evidence of chronic inflammation in veterans with GWI has emerged from previous observational studies. The goal of this trial is to determine if reducing the GWI-associated chronic inflammation is an effective treatment for GWI. This is a randomized, two group, placebo controlled, double blind clinical trial. The treatment group will receive a low dose (2x5mg) once a day of delayed-release prednisone (Rayos) for 8 weeks. The placebo group will receive matching placebo (2x5mg) once a day for 8 weeks. The primary outcome measure for this clinical trial is a change from baseline of HRQOL with respect to physical functioning and symptoms. The secondary outcome measures include changes from baseline of peripheral blood levels of GWI-associated biomarkers of inflammation, changes from baseline of GWI-associated symptoms (chronic pain, fatigue, and cognitive impairment), and a change from baseline of HRQOL with respect to mental functioning.

ELIGIBILITY:
Inclusion Criteria:

* Scores moderate-severe on at least 3 out of 6 domains from the Kansas GWI Case Definition
* Deployed, (and honorably discharged), from the Kuwaiti Theater of Operation (August 2, 1990-July 31, 1991)

Exclusion Criteria:

* Hospitalization anytime since 1990 for Alcohol or Drug Dependence, Depression, or PTSD
* Known hypersensitivity to Prednisone
* Liver, (active or recent Hepatitis B or C treatment with a completion date within the past 6 months, or alcohol liver disease), or Kidney Disease (Hep B and C ok if after 6 months of treatment)
* Treated Diabetes
* Females who are Pregnant or Nursing
* Female who refuses to use an accepted method of birth control
* Exclusionary Labs: C-Reactive Protein >25, Creatinine Clearance <30, EFGR ≥ 30, Hgb A1-C >7, Glucose >120, WBC >12, RBC >6.2, Hematocrit >60, Hemoglobin <11, Platelets <100, Liver Function Tests (2 x the upper limit of AST and ALT, 2 x the upper limit of Total Bilirubin, and Alkaline Phosphatase)
* Has Inflammatory Arthritis (RA, or Psoriatic Arthritis, Spondylitis, Polyarthritis)
* Reactive Arthritis, or IBD associated Arthritis
* Has any major inflammatory disease (acute Chronic Infections, Ulcerative Colitis, Crohn's Disease, Inflammatory lung diseases- COPD or Asthma requiring steroid treatment, Pericarditis, Vasculitis)
* Has an chronic/active infection
* Chronic use of Prednisone or Corticosteroids (occasional inhaled use of steroids acceptable)
* Active Gum Disease or Dental Infection
* Has been diagnosed with Lupus, Stroke, or Multiple Sclerosis. or any other diagnosis that produces symptoms of fatigue, cognitive impairment, or pain will be excluded based on the Kansas GWI Case definition
* Has a condition that may interfere with the ability to accurately report symptoms, (Severe Psychiatric Problems, Schizophrenia, Bipolar Disorder, Alcohol or Drug Dependence requiring hospitalization, or regular illegal drug use)
* Heart Disease (other than Hypertension), Heart Failure or Coronary Heart Disease requiring hospitalization within the past 12 months
* Cancer (other than basal cell skin cancer), requiring treatment within the past 12 months, or life expectancy of less than 1 year.
* Hospitalization within the past 3 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2015-07; Primary Completion 2023-10-19 (Actual); Study Completion 2023-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald R Bach, PhD, Principal Investigator — Minneapolis Veterans Affairs Medical Center
Locations (1):
- Minneapolis Veterans Affairs Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
After publication, all deidentified study data will be made available to other investigators upon request. Data sharing rule of the journal will apply.
Supporting Information: Study Protocol, ICF
Time Frame: After publication for as long as specified by the journal
Access Criteria: Established investigators with legitimate scientific credentials

REFERENCES:
- [Background] Bach RR, Rudquist RR. Gulf war illness inflammation reduction trial: A phase 2 randomized controlled trial of low-dose prednisone chronotherapy, effects on health-related quality of life. PLoS One. 2023 Jun 15;18(6):e0286817. doi: 10.1371/journal.pone.0286817. eCollection 2023. PMID 37319244
- See also: link to citation — http://journals.plos.org/plosone/article?id=10.1371/journal.pone.0286817

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Modified-Release Prednisone | Placebo
Started | 42 | 41
Completed | 41 | 40
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Modified-Release Prednisone | Placebo | Total
Number analyzed (Participants) | 42 | 41 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 41 | 83
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (4.0) | 52.2 (6.4) | 51.0 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 40 | 38 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 41 | 40 | 81
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 39 | 38 | 77
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 42 | 41 | 83

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of Veterans RAND 36-Item Health Survey Physical Component Summary Score (PCS) Scores at 8 and 16 Weeks
Description: The SF-36V is a modification of the well-established Medical Outcomes Study Short Form Health Survey (SF-36). It surveys eight concepts of health: physical functioning, role limitations because of physical problems, bodily pain, general health perceptions, energy/vitality, social functioning, role limitations due to emotional problems and mental health. From these concepts, two summary component scores are derived: a Physical Component Summary (PCS) and a Mental Component Summary (MCS).
  To calculate PCS, scales are standardized with a scoring algorithm or by the scoring software. Scores are standardized and range from 0 to 100, with a US population mean of 50 points and a SD of 10 points. The PCS and the MCS have been demonstrated to have excellent psychometric properties. SF-36V PCS is a measure of HRQOL with respect to physical functioning and symptoms. Higher scores indicate better health status,
Time Frame: 0, 8, and 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Modified-Release Prednisone | Placebo
Number analyzed (Participants) | 42 | 41
units on a scale
  baseline | 40.8 (9.2) | 41.5 (9.9)
  8 weeks | 43.5 (9.6) | 43.4 (9.8)
  16 weeks | 40.8 (8.3) | 41.4 (10.8)

2. Secondary Outcome: Change From Baseline of McGill Pain Questionnaire-short Form (MPQ) Scores at 8 and 16 Weeks
Description: MPQ asks questions about sensory pain, affective pain, pain now, and typical pain
Time Frame: 0, 8, and 16 weeks
Reporting Status: Not Posted, anticipated posting 2026-01

3. Secondary Outcome: Change From Baseline of Multidimensional Fatigue Inventory (MFI) Scores at 8 and 16 Weeks
Description: MFI asks questions about general fatigue, physical fatigue, reduced activity, reduced motivation, and mental fatigue.
Time Frame: 0, 8, and 16 weeks
Reporting Status: Not Posted, anticipated posting 2026-01

4. Secondary Outcome: Change From Baseline of Cognitive Failures Questionnaire (CFQ) Scores at 8 and 16 Weeks
Description: CFQ asks questions about cognitive symptoms such as attention, concentration, and memory
Time Frame: 0, 8, and 16 weeks
Reporting Status: Not Posted, anticipated posting 2026-01

5. Secondary Outcome: Change From Baseline of Veterans RAND 36-Item Health Survey Mental Component Summary Score (MCS) Scores at 8 and 16 Weeks
Description: SF-36V MCS is a measure of HRQOL with respect to mental functioning. The SF-36V is a modification of the well-established Medical Outcomes Study Short Form Health Survey (SF-36). It surveys eight concepts of health: physical functioning, role limitations because of physical problems, bodily pain, general health perceptions, energy/vitality, social functioning, role limitations due to emotional problems and mental health. From these concepts, two summary component scores are derived: a Physical Component Summary (PCS) and a Mental Component Summary (MCS).
  To calculate MCS, scales are standardized with a scoring algorithm or by the scoring software. Scores are standardized and range from 0 to 100, with a US population mean of 50 points and a SD of 10 points. The PCS and the MCS have been demonstrated to have excellent psychometric properties. SF-36V MCS is a measure of HRQOL with respect to mental functioning and symptoms. Higher scores indicate better health status,
Time Frame: 0, 8, and 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Modified-Release Prednisone | Placebo
Number analyzed (Participants) | 42 | 41
units on a scale
  baseline | 40.8 (13.3) | 40.4 (12.8)
  8 weeks | 42.4 (13.2) | 43.1 (11.9)
  16 weeks | 40.1 (13.2) | 42.7 (12.0)

6. Secondary Outcome: Change From Baseline of Gulf War Illness-associated Peripheral Blood Biomarkers
Description: Peripheral blood biomarker levels are quantified by multi-analyte profiling (MAP) and complete blood count (CBC) analyses
Time Frame: 0, 8, and 16 weeks
Reporting Status: Not Posted, anticipated posting 2026-01

ADVERSE EVENTS:
Time Frame: 16 weeks
Groups:
- Treatment: 2x5mg MR-prednisone QD at bedtime
- Placebo: 2 matching placebo tablets QD at bedtime
Arm/Group | Treatment | Placebo
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/41
Other Adverse Events (participants affected / at risk) | 0/42 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2013-09-12): https://cdn.clinicaltrials.gov/large-docs/92/NCT02506192/Prot_SAP_000.pdf
  • Informed Consent Form (2015-10-05): https://cdn.clinicaltrials.gov/large-docs/92/NCT02506192/ICF_001.pdf